CLINICAL TRIAL: NCT04620252
Title: Enhancing the Fluoride Retention in the Mouth by Chewing a Calcium Supplement Before Fluoride Rinse
Brief Title: Effect of Chewing a Calcium Supplement Before Fluoride Rinse on Salivary Fluoride
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Livia Tenuta, DDS, MS, PhD, Associate Professor, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: HUM00176242
Record Dates: First submitted 2020-11-05; First posted 2020-11-06 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chewing calcium supplements (Experimental): Participants were given one of 4 different treatments to chew: a negative control group and 3 calcium supplements with different calcium compositions.
  Participants were randomized to determine the sequence of exposure to the different treatments.
  Interventions: Drug: Inactive supplement; Drug: Tricalcium phosphate supplement; Drug: Calcium carbonate supplement; Drug: Calcium citrate supplement
- Fluoride rinse (Experimental): Participants rinsed with an over the counter sodium fluoride rinse for 1 min, after having chewed a candy (negative control), a calcium calcium carbonate or a calcium citrate supplement.
  Interventions: Drug: Inactive supplement and fluoride mouthwash; Drug: Calcium carbonate supplement and fluoride mouthwash; Drug: Calcium citrate supplement and fluoride mouthwash

INTERVENTIONS:
Drug: Inactive supplement — Chewable candy (negative control), chewed for 30 seconds.
  Arms: Chewing calcium supplements
Drug: Tricalcium phosphate supplement — Chewable tricalcium phosphate supplement, chewed for 30 seconds.
  Arms: Chewing calcium supplements
Drug: Calcium carbonate supplement — Chewable calcium carbonate supplement, chewed for 30 seconds.
  Arms: Chewing calcium supplements
Drug: Calcium citrate supplement — Chewable calcium citrate supplement, chewed for 30 seconds.
  Arms: Chewing calcium supplements
Drug: Inactive supplement and fluoride mouthwash — A chewable candy chewed for 30 seconds, immediately followed by a 1 minute rinse with an over the counter sodium fluoride mouthwash, at a concentration of 0.05% (226 parts per millim (ppm) of fluoride).
  Arms: Fluoride rinse
Drug: Calcium carbonate supplement and fluoride mouthwash — A calcium carbonate supplement chewed for 30 seconds, immediately followed by a 1 minute rinse with an over the counter sodium fluoride mouthwash, at a concentration of 0.05% (226 parts per millim (ppm) of fluoride).
  Arms: Fluoride rinse
Drug: Calcium citrate supplement and fluoride mouthwash — A calcium citrate supplement chewed for 30 seconds, immediately followed by a 1 minute rinse with an over the counter sodium fluoride mouthwash, at a concentration of 0.05% (226 parts per millim (ppm) of fluoride).
  Arms: Fluoride rinse

SUMMARY:
The anticaries effect of fluoride is through the increase in fluoride presence and retention in the oral fluids, reducing dental demineralization and enhancing remineralization. Previous studies showed that a preapplication of calcium (in a rinse) prior to administration of fluoride greatly enhances fluoride concentration in the mouth and the anticaries effect of fluoride. The hypothesis of this study is that the same can be achieved by chewing a calcium supplement prior to a fluoride rinse. The first goal is to determine if chewing these calcium supplements will increase calcium concentration in the oral fluids above baseline levels. Secondly, the calcium supplement with the highest calcium release will be tested before a fluoride rinse to assess the increased retention of fluoride in the oral fluids when compared with the fluoride rinse alone. In both parts, healthy volunteers will participate and saliva will be collected to assess calcium and fluoride concentration.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Reported good general health
* Reported good oral health
* Having at least 20 teeth in the mouth, being at least 4 (natural or crowned) teeth in all four quadrants of the mouth
* Having normal salivary flow rate according to direct flow rate determination methods
* Agreement to adhere to the study protocol

Exclusion Criteria:

* Unable to understand and/or follow study instructions
* Hyposalivation
* Active periodontitis, identified by frequent bleeding of the gums
* Oral pain
* In need of urgent dental care

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Calcium concentration in saliva at baseline | Baseline
  Saliva collected as one spit, immediately before chewing one of the calcium supplements to be tested in Arm 1. Calcium concentration determined using a colorimetric method.
Calcium concentration in the mixture of saliva and chewed calcium supplement | Immediately after the 30-second chewing of calcium supplement
  Saliva and remnants of the chewed calcium supplement collected at the end of the chewing period (30 seconds) in Arm 1. Calcium concentration determined using a colorimetric method.
Calcium concentration in saliva at 15 seconds | 15 seconds after chewing calcium supplement
  Saliva collected as one spit, 15 seconds after chewing the calcium supplement in Arm 1. Calcium concentration determined using a colorimetric method.
Calcium concentration in saliva at 30 seconds | 30 seconds after chewing calcium supplement
  Saliva collected as one spit, 30 seconds after chewing the calcium supplement in Arm 1. Calcium concentration determined using a colorimetric method.
Calcium concentration in saliva at 45 seconds | 45 seconds after chewing calcium supplement
  Saliva collected as one spit, 45 seconds after chewing the calcium supplement in Arm 1. Calcium concentration determined using a colorimetric method.
Calcium concentration in saliva at 60 seconds | 60 seconds after chewing calcium supplement
  Saliva collected as one spit, 60 seconds after chewing the calcium supplement in Arm 1. Calcium concentration determined using a colorimetric method.
Calcium concentration in saliva at 120 seconds | 120 seconds after chewing calcium supplement
  Saliva collected as one spit, 120 seconds after chewing the calcium supplement in Arm 1. Calcium concentration determined using a colorimetric method.
Calcium concentration in saliva at 180 seconds | 180 seconds after chewing calcium supplement
  Saliva collected as one spit, 180 seconds after chewing the calcium supplement in Arm 1. Calcium concentration determined using a colorimetric method.
Calcium concentration in saliva at 240 seconds | 240 seconds after chewing calcium supplement
  Saliva collected as one spit, 240 seconds after chewing the calcium supplement in Arm 1. Calcium concentration determined using a colorimetric method.
Calcium concentration in saliva at 300 seconds | 300 seconds after chewing calcium supplement
  Saliva collected as one spit, 300 seconds after chewing the calcium supplement in Arm 1. Calcium concentration determined using a colorimetric method.
Area under the curve of calcium concentration in saliva | Baseline, 15, 30, 45, 60, 120, 180, 240 and 300 seconds after chewing calcium supplements
  Calcium concentration in saliva collected at baseline (before chewing the supplements), and 15, 30, 45, 60, 120, 180, 240 and 300 seconds after chewing the supplements in Arm 1 expressed as the area under the curve of calcium concentration in saliva as a function of time (milimolar x min).
Fluoride concentration in saliva at baseline | Baseline
  Saliva will be collected for 2 min, immediately before chewing a calcium supplement and/or rinse with the fluoride mouthrinse in Arm 2. Fluoride concentration will be determined using an ion-specific electrode.
Fluoride concentration in saliva at time 0 | 0 minutes after chewing supplement/mouthwashing
  Saliva and remnants of the fluoride mouth rinse collected at the end of the rinsing period (1 minute) in Arm 2. Fluoride concentration determined using an ion-specific electrode.
Fluoride concentration in saliva at 5 min | 5 minutes after chewing supplement/mouthwashing
  Saliva will be collected for 2 min, 5 min after chewing a calcium supplement and/or rinse with the fluoride mouthrinse in Arm 2. Fluoride concentration will be determined using an ion-specific electrode.
Fluoride concentration in saliva at 15 min | 15 minutes after chewing supplement/mouthwashing
  Saliva collected for 2 min, 15 min after chewing a calcium supplement and/or rinse with the fluoride mouthrinse in Arm 2. Fluoride concentration determined using an ion-specific electrode.
Fluoride concentration in saliva at 30 min | 30 minutes after chewing supplement/mouthwashing
  Saliva collected for 2 min, 30 min after chewing a calcium supplement and/or rinse with the fluoride mouthrinse in Arm 2. Fluoride concentration determined using an ion-specific electrode.
Fluoride concentration in saliva at 60 min | 60 minutes after chewing supplement/mouthwashing
  Saliva collected for 2 min, 60 min after chewing a calcium supplement and/or rinse with the fluoride mouthrinse in Arm 2. Fluoride concentration determined using an ion-specific electrode.
Fluoride concentration in saliva at 120 min | 120 minutes after chewing supplement/mouthwashing
  Saliva collected for 2 min, 120 min after chewing a calcium supplement and/or rinse with the fluoride mouthrinse in Arm 2. Fluoride concentration determined using an ion-specific electrode.
Area under the curve of fluoride concentration in saliva | Baseline, 5, 15, 30, 60 and 120 minutes after chewing supplement/mouthwashing
  Fluoride concentration in saliva collected at baseline (before treatments), and 0, 5, 15, 30, 60 and 120 minutes after chewing the supplements and/or rinsing the fluoride mouthrinse in Arm 2 expressed as the area under the curve of fluoride concentration in saliva as a function of time (micromolar x min).

CONTACTS AND LOCATIONS:
Overall Officials: Livia M Tenuta, DDS, MS, PhD, Principal Investigator — Associate Professor, University of Michigan
Locations (1):
- School of Dentistry, University of Michigan, Ann Arbor, Michigan, United States